CLINICAL TRIAL: NCT02036125
Title: Syndrome du Tunnel Carpien - Essai Clinique randomisé évaluant l'efficacité de l'Utilisation de l'échographie Lors de l'Infiltration de corticostéroïdes
Brief Title: Carpal Tunnel Syndrome - Randomized Clinical Trial Evaluating Effectiveness of Ultrasound in Corticosteroid Injection
Acronym: STC-EI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Alessandra Bruns, MD, FRCPC, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-143
Record Dates: First submitted 2014-01-11; First posted 2014-01-14 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Corticosteroid; Ultrasound; Guided injection
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Ultrasonography; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound guided injection (Experimental): Ultrasound guided injection of 40 mg of methylprednisolone
  Interventions: Device: Ultrasound; Drug: methylprednisolone
- Blind injection (Active Comparator): Blind injection of 40 mg of methylprednisolone
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Device: Ultrasound — Subjects will receive an ultrasound guided injection of 40 mg of methylprednisolone.
  Arms: Ultrasound guided injection
Drug: methylprednisolone — Subjects will receive a blind injection of 40 mg of methylprednisolone.

SUMMARY:
The objective of this study is to evaluate the efficacy of ultrasound guided corticosteroid injection in reducing symptoms caused by carpal tunnel syndrome.

DETAILED DESCRIPTION:
Corticosteroid injection is routinely given for treating carpal tunnel syndrome. The objective of this study is to evaluate the efficacy of ultrasound guided corticosteroid injection in reducing symptoms caused by carpal tunnel syndrome.

In this randomised clinical trial, 50 patients with both a clinical and electromyographic diagnosis of mild to moderate carpal tunnel syndrome will be recruited from the Centre Hospitalier Universitaire de Sherbrooke (CHUS). Subjects will be randomised to ultrasound guided or blind injection groups. All subjects will receive 40 mg of methylprednisolone. The primary outcome will be the Boston Carpal Tunnel Syndrome Questionnaire - Symptom Severity Scale at baseline and 3 months post injection. Both subjects and assessors will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65
* Understanding written and spoken french
* Diagnostic of carpal tunnel syndrome : Classic of probable based on the Katz Hand Diagram and mild to moderate based on the electrodiagnosis studies

Exclusion Criteria:

* Carpal tunnel injection in the last 6 months
* Constant symptoms in medial nerve area
* Thenar eminence atrophy
* Absolute contraindication to corticosteroid injection : infective arthritis, bacterial endocarditis, local cellulitis of skin infection, coagulopathy, corticosteroid or latex allergy
* Secondary diagnosis based on the ultrasound : arthrosynovial cyst, flexor tenosynovitis, ganglion
* Known cognitive disorder
* Anticoagulant therapy
* Diseases known to cause carpal tunnel syndrome : Diabetes mellitus, hypothyroidism, connective tissue disease, rheumatic disease and moderate or severe chronic renal impairment
* Radiculopathy
* Polyneuropathy
* Pregnancy
* Ancient ipsilateral wrist fracture
* Ancient ipsilateral wrist surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire - Symptom Severity Scale | 3 months
  The Boston Questionnaire is self-applied by the patient. It has a symptom severity scale and a functional status scale.

SECONDARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire - Functional Status Scale | 3 months
  The Boston Questionnaire is self-applied by the patient. It has a symptom severity scale and a functional status scale.
DASH questionnaire | 3 months
Numeric Pain Rating Scale | 3 months
  Mean pain felt in the last 2 weeks
Ultrasound measured medial nerve area in carpal tunnel | 3 months
Ultrasound measured medial nerve area difference between pronator quadratus and carpal tunnel | 3 months
Ultrasound hypervascularisation of medial nerve in carpal tunnel | 3 months
Numeric Pain Rating Scale | Baseline
  Pain during injection
Global Rating of Change | 3 months
  The Global Rating of Change scale is meant to quantify the improvement or deterioration perceived by the patient.

OTHER OUTCOMES:
Trial group assignment - Patient | 3 months
  Questionnaire to verify patient's beliefs regarding his group allocation at follow-up.
Trial group assignment - Assessor | 3 months
  Questionnaire to verify assessor's beliefs regarding a patient group allocation at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Bruns, Md, FRCPC, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada